CLINICAL TRIAL: NCT04613115
Title: Study on the Relationship Between Variations in the Branching Pattern of the Main Arteries and Patency of Arteriovenous Fistulae in the Upper Limb
Brief Title: Relationship Between Arterial Variations and Patency of Arteriovenous Fistulae
Status: Completed | Type: Observational
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TRECKY2020-101
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2020-10

CONDITIONS: Arteriovenous Fistula; Ultrasound; Artery
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: patients without uremia and variant arteries
- Group B: patients without uremia, but with variant arteries
- Group C: patients with uremia ,without variant arteries
- Group D: patients with uremia and variant arteries

SUMMARY:
In 2019, KDOQI considered that uremic patients with a life expectancy of more than one year should require hemodialysis as an effective renal replacement therapy before preparation of kidney transplantation. Arteriovenous fistula, as the lifeline of uremic patients, plays an important role in their daily hemodialysis. The patency of arteriovenous fistula is largely restricted by the inflow artery. According to available medical literatures, an incidence rate of variations in the branching pattern of the main arteries in the upper limb is ranged from 7.2% to 25.0%. and there is a large difference in the incidence rate between sex and race, furthermore, the incidence rate of variations in the branching pattern of the main arteries in the upper limb of Chinese is still unclear. The brachial artery is the main artery of the upper limb. It gives off two terminal branches at the distal end of the elbow crease, the radial and ulnar arteries, the former one often serves as an arterial inflow to create an arteriovenous fistula in the forearm. High bifurcation of the brachial artery (HBBA) seems to be a common variation which may result in immaturity or disfunction of arteriovenous fistulas. Therefore, the purpose of this study is to investigate the variations in the branching pattern of the main arteries in the upper limb of Chinese, in order to study on the hemodynamic changes, and their influence on the establishment, maturation and failure of arteriovenous fistulas in the upper limb.

DETAILED DESCRIPTION:
This is a prospective analysis research, collecting information after patients admission, including basic information, primary disease status, dialysis intubation status, current dialysis access status, last dialysis access maintenance status and other relevant data. The above-mentioned information data is collected when the patient is admitted into the department of vascular surgery, and is recorded in the "Information Collection, Diagnosis and Treatment Process of Hemodialysis Patients in the Department of Vascular Surgery" form for retention and filing.

During the study period, all patients who were admitted to the vascular surgical department and signed the "Informed Consent" before the upper extremity artery screening according to the corresponding procedures.

ELIGIBILITY:
Inclusion Criteria:

* patients of vascular surgical Inpatient department
* patients will sign the "Informed Consent" and be able to receive related ultrasound examinations

Exclusion Criteria:

* Patients of other surgical Inpatient department

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: all patients who were admitted to the vascular surgical Inpatient department from outpatient department.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
the variations in the branching pattern of the main arteries in the upper limb of Chinese. | baseline
  brachio-radial artery、superficial brachio-radial artery、brachio-ulnar artery、superficial brachio-ulnar artery、brachioulnoradial artery、brachiointerosseous artery.
Patency of arteriovenous fistulae in the upper limb | 1 year
  functional patency、primary patency、primary assisted patency、secondary patency

CONTACTS AND LOCATIONS:
Overall Officials: ZhengYa Yu, MD, Study Director — Department of Vascular Surgery, Beijing Tongren Hospital, Capital Medical University.; Xin Chen, MM, Principal Investigator — Department of Vascular Surgery, Beijing Tongren Hospital, Capital Medical University.
Locations (1):
- Department of Vascular Surgery, Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] KEEN JA. A study of the arterial variations in the limbs, with special reference to symmetry of vascular patterns. Am J Anat. 1961 May;108:245-61. doi: 10.1002/aja.1001080303. No abstract available. PMID 14454801
- [Background] Tsoucalas G, Eleftheriou A, Panagouli E. High Bifurcation of the Brachial Artery: An Embryological Overview. Cureus. 2020 Feb 25;12(2):e7097. doi: 10.7759/cureus.7097. PMID 32231893
- [Background] Aragao JA, da Silva AC, Anunciacao CB, Reis FP. Median artery of the forearm in human fetuses in northeastern Brazil: anatomical study and review of the literature. Anat Sci Int. 2017 Jan;92(1):107-111. doi: 10.1007/s12565-015-0322-x. Epub 2016 Jan 8. PMID 26747631
- [Background] Cikla U, Mukherjee D, Tumturk A, Baskaya MK. Overcoming End-to-End Vessel Mismatch During Superficial Temporal Artery-Radial Artery-M2 Interposition Grafting for Cerebral Ischemia: Tapering Technique. World Neurosurg. 2018 Feb;110:85. doi: 10.1016/j.wneu.2017.10.162. Epub 2017 Nov 6. PMID 29122732
- [Background] Jennings WC, Mallios A, Mushtaq N. Proximal radial artery arteriovenous fistula for hemodialysis vascular access. J Vasc Surg. 2018 Jan;67(1):244-253. doi: 10.1016/j.jvs.2017.06.114. Epub 2017 Sep 11. PMID 28912005
- [Background] Kachlik D, Hajek P, Konarik M, Krchov M, Baca V. Coincidence of superficial brachiomedian artery and bitendinous palmaris longus: a case report. Surg Radiol Anat. 2016 Jan;38(1):147-51. doi: 10.1007/s00276-015-1512-x. Epub 2015 Jul 2. PMID 26134151
- [Background] Shetty SD, Nayak B S, Madhav N V, Sirasanagandla SR, P A. The abnormal origin, course and the distribution of the arteries of the upper limb: a case report. J Clin Diagn Res. 2012 Oct;6(8):1414-6. doi: 10.7860/JCDR/2012/4183.2373. PMID 23205361
- [Background] Singer G, Marterer R, Till H, Schmidt B. A rare anatomic variation of the superficial palmar branch of the radial artery causing pain. Surg Radiol Anat. 2018 Mar;40(3):349-352. doi: 10.1007/s00276-017-1936-6. Epub 2017 Nov 9. PMID 29124345
- [Background] Lee H, Moon YS, Park HS, Kim HT, Choi IJ. A radial artery originating from the thoracoacromial artery. Surg Radiol Anat. 2016 Jul;38(5):631-3. doi: 10.1007/s00276-015-1576-7. Epub 2015 Oct 22. PMID 26493986
- [Background] Nasr AY. The radial artery and its variations: anatomical study and clinical implications. Folia Morphol (Warsz). 2012 Nov;71(4):252-62. PMID 23197145
- [Background] Wysiadecki G, Polguj M, Haladaj R, Topol M. Low origin of the radial artery: a case study including a review of literature and proposal of an embryological explanation. Anat Sci Int. 2017 Mar;92(2):293-298. doi: 10.1007/s12565-016-0371-9. Epub 2016 Sep 15. PMID 27631096
- [Background] Hamahata A, Nakazawa H, Takeuchi M, Sakurai H. Usefulness of radial recurrent artery in transplant of radial forearm flap: an anatomical and clinical study. J Reconstr Microsurg. 2012 Mar;28(3):195-8. doi: 10.1055/s-0031-1301071. Epub 2012 Jan 24. PMID 22274767
- [Background] Vazquez T, Sanudo JR, Carretero J, Parkin I, Rodriguez-Niedenfuhr M. Variations of the radial recurrent artery of clinical interest. Surg Radiol Anat. 2013 Oct;35(8):689-94. doi: 10.1007/s00276-013-1094-4. Epub 2013 Feb 26. PMID 23440497
- [Background] Rodriguez-Niedenfuhr M, Vazquez T, Nearn L, Ferreira B, Parkin I, Sanudo JR. Variations of the arterial pattern in the upper limb revisited: a morphological and statistical study, with a review of the literature. J Anat. 2001 Nov;199(Pt 5):547-66. doi: 10.1046/j.1469-7580.2001.19950547.x. PMID 11760886
- [Background] Lioupis C, Mistry H, Junghans C, Haughey N, Freedman B, Tyrrell M, Valenti D. High brachial artery bifurcation is associated with failure of brachio-cephalic autologous arteriovenous fistulae. J Vasc Access. 2010 Apr-Jun;11(2):132-7. doi: 10.1177/112972981001100209. PMID 20155716
- [Background] Kirksey L. Unrecognized high brachial artery bifurcation is associated with higher rate of dialysis access failure. Semin Dial. 2011 Nov-Dec;24(6):698-702. doi: 10.1111/j.1525-139X.2011.00923.x. Epub 2011 Sep 4. PMID 21895770 (Retraction: PMID 28251695 Semin Dial. 2017 Mar;30(2):183)
- [Background] Beathard GA, Lok CE, Glickman MH, Al-Jaishi AA, Bednarski D, Cull DL, Lawson JH, Lee TC, Niyyar VD, Syracuse D, Trerotola SO, Roy-Chaudhury P, Shenoy S, Underwood M, Wasse H, Woo K, Yuo TH, Huber TS. Definitions and End Points for Interventional Studies for Arteriovenous Dialysis Access. Clin J Am Soc Nephrol. 2018 Mar 7;13(3):501-512. doi: 10.2215/CJN.11531116. Epub 2017 Jul 20. PMID 28729383
- [Background] Yang HJ, Gil YC, Jung WS, Lee HY. Variations of the superficial brachial artery in Korean cadavers. J Korean Med Sci. 2008 Oct;23(5):884-7. doi: 10.3346/jkms.2008.23.5.884. PMID 18955798
- [Background] Pham XD, Kim JJ, Parrish AB, Tom C, Ihenachor EJ, Mina D, de Virgilio C. Racial and Gender Differences in Arterial Anatomy of the Arm. Am Surg. 2016 Oct;82(10):973-976. PMID 27779986